CLINICAL TRIAL: NCT03400046
Title: The Correlation Between Nutritional Support Regimens and Muscle Mass in Patients With Chronic Intestinal Failure
Brief Title: The Correlation Between Nutrients and Muscle Mass
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Department General surgery, Jinling Hospital, China
Other Study IDs: 201502022-4
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Nutritional Support; Muscle Loss
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nutritional Product Supplementation — Patients with chronic intestinal failure were administered nutritional support including enteral and parenteral nutrition.

SUMMARY:
Patients who are suffer from CIF often develop muscle wasting because of hypercatabolism.The relationship between different nutrition support formulas and lean body mass is still unclear. The purpose of this study is to investigate the relationship between nutrition support and muscle mass and attempt to find the nutrients which will benefit lean body mass in patients with CIF.

DETAILED DESCRIPTION:
Chronic intestinal failure (CIF) is defined as the malabsorption and nutrients deficiency mainly caused by severe gastrointestinal benign diseases such as intestinal ﬁstula, short bowel, and mechanical obstruction and some malignant diseases such as end-stage intra-abdominal or pelvic cancers . CIF is one of the rarest of organ failures all over the world and patients suffer from CIF often requires a prolonged time to recover . Hypercatabolism caused by diseases stress, inflammation and reduced nutrient intake indicates that patients with CIF need long-term nutritional support .

Patients who are suffer from CIF often develop muscle wasting because of hypercatabolism. Moreover, studies showed that low muscle mass and muscle wasting during critical illness are associated with poor clinical outcomes and hampered rehabilitation. Except Resistance training, sufficient nutrients supplement also play important roles in maintaining the skeletal muscle mass. Guidelines recommended that nutritional support regimens in patients should be individualized and adjusted over time based on formal nutritional assessment . However, almost all guidelines only recommended the total energy and protein requirements based on the results of basal metabolic rate (BMR) and nitrogen balance rather than the lean body mass . The relationship between different nutrition support formulas and lean body mass is still unclear.

The purpose of this study is to investigate the relationship between nutrition support and muscle mass and attempt to find the nutrients which will benefit lean body mass in patients with CIF.

All adult CIF patients (age ≥18 years) receiving nutrition support were included. The exclusion criteria were hepatic insufficiency (alanine transaminase/aspartate transaminase ratio 200% above normal range or bilirubin >3 mg/dL), renal insufficiency (serum creatinine [Scr] >1.5 mg/dL), acute or life-threatening diseases (e.g., shock, collapse, stroke, coma of unknown etiology, or recent cardiac infarction), and pregnant or breast-feeding women. The study was approved by the ethics committee of Jinling Hospital, Medical School of Nanjing University.

The lean body mass include soft lean mass (SLM), skeletal muscle mass (SMM) and fat free mass (FFM) which were measured and recorded by body composition analyzer (InBody S10, Biospace) at the time of admission and discharge respectively.The deviation of lean body mass was calculated by the difference between admission and discharge, and then symbolized as ∆SLM, ∆SMM and ∆FFM. Basic and nutritional information of CIF patients was measured weekly after hospital admission, including age, sex, BMI, NRS-2002 score, SGA grade, etiology of malnutrition, daily energy & protein intake via EN & PN.

ELIGIBILITY:
Inclusion Criteria:

- All adult CIF patients (age ≥18 years) receiving nutrition support were included

Exclusion Criteria:

- Hepatic insufficiency (alanine transaminase/aspartate transaminase ratio 200% above normal range or bilirubin >3 mg/dL), renal insufficiency (serum creatinine [Scr] >1.5 mg/dL), acute or life-threatening diseases (e.g., shock, collapse, stroke, coma of unknown etiology, or recent cardiac infarction), and pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a single clinical nutrition center of a tertiary referral hospital in China to investigate the relationship between nutrients and muscle mass in CIF patients. The data used were accumulated at the center between September 2013 and September 2017.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Body composition | From date of patients enrollment until the date of patients discharge from hospital, assessed up to 2 months.
  soft lean mass/skeletal muscle mass/fat free mass

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [1] Bielawska B, Allard JP: Parenteral Nutrition and Intestinal Failure. Nutrients 2017, 9. [2] Pironi L, Arends J, Bozzetti F, Cuerda C, Gillanders L, Jeppesen PB, Joly F, Kelly D, Lal S, Staun M, Szczepanek K, Van Gossum A, Wanten G, Schneider SM: ESPEN guidelines on chronic intestinal failure in adults. Clinical nutrition 2016, 35:247-307. [3] Pironi L: Definitions of intestinal failure and the short bowel syndrome. Best Pract Res Clin Gastroenterol 2016, 30:173-85. [4] Feinberg J, Nielsen EE, Korang SK, Halberg Engell K, Nielsen MS, Zhang K, Didriksen M, Lund L, Lindahl N, Hallum S, Liang N, Xiong W, Yang X, Brunsgaard P, Garioud A, Safi S, Lindschou J, Kondrup J, Gluud C, Jakobsen JC: Nutrition support in hospitalised adults at nutritional risk. The Cochrane database of systematic reviews 2017, 5:Cd011598. [5] Taylor BE, McClave SA, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C, Society of Critical Care M, the American Society of P, Enteral N: Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). Crit Care Med 2016, 44:390-438. [6] McClave SA, DiBaise JK, Mullin GE, Martindale RG: ACG Clinical Guideline: Nutrition Therapy in the Adult Hospitalized Patient. Am J Gastroenterol 2016, 111:315-34.